CLINICAL TRIAL: NCT05947201
Title: Neoadjuvant Treatment of Cadonilimab Combined Albumin-paclitaxel, Cisplatin and Fluorouracil for Resectable Locally Advanced Esophageal Squamous Cell Carcinoma：A Single-Arm Phase 2 Clinical Trial
Brief Title: Neoadjuvant Treatment of Cadonilimab Combined Albumin-paclitaxel, Cisplatin and Fluorouracil for Resectable Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weijia Fang, MD (Other)
Collaborators: Akeso Pharmaceuticals, Inc. (Other)
Responsible Party: Sponsor-Investigator, Weijia Fang, MD, Oncology Department director, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPITAL
Record Dates: First submitted 2023-05-07; First posted 2023-07-17 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: The Efficacy and Safety of Therapy Efficacy for Locally Advanced ESCC
MeSH Terms: interventions — Cisplatin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: Patients fulfilling Eligibility Criteria will be included in our study. ESCC participants in this study will be given intravenous administration of AK104 (10 mg/kg d1) combined with cisplatin (20 mg/m2 on d1-3) and albumin paclitaxel (100mg/m2 on d1, d8), fluorouracil (600 mg/m2 on d1-5) every three weeks for a cycle of treatment, which will be conducted two or three cycles, and radical surgery within 4-6 weeks after the last administration. Treatments will be administrated until disease progression, unacceptable adverse events (AE), concomitant diseases that hinder continued treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AK104+cisplatin+albumin paclitaxel+fluorouracil (Experimental): AK104 (10 mg/kg d1), in combination with cisplatin (20 mg/m2 on d1-3) and albumin paclitaxel (100mg/m2 on d1,d8), fluorouracil (600 mg/m2 on d1-5) Q3W, intravenously
  Interventions: Drug: Cadonilimab Combined Albumin-paclitaxel, Cisplatin and Fluorouracil

INTERVENTIONS:
Drug: Cadonilimab Combined Albumin-paclitaxel, Cisplatin and Fluorouracil — If the addition of Cadonilimab to neoadjuvant chemotherapy further improve the efficiency for locally advanced esophageal squamous cell carcinoma
  Other Names: rutine

SUMMARY:
This is a single-arm clinical study to evaluate the efficacy and safety of Cadonilimab in combination with preoperative chemotherapy for locally advanced esophageal squamous cell carcinoma Locally Advanced Esophageal Squamous Cell Carcinoma

DETAILED DESCRIPTION:
Esophageal cancer is the eighth most lethal tumor and the sixth leading cause of cancer-related deaths worldwide. Esophageal squamous cell carcinoma accounts for up to 95% of the pathological types and threatens the health of chinese residents. Investigator designed a single-arm, open-label, phase II trial and the purpose of this study is to observe and evaluate the efficacy and safety of Cadonilimab combined with preoperative chemotherapy for locally advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have given their consent and signed an informed consent form, are willing and able to comply with the study visits, treatment, laboratory tests, and other trial procedures.
2. Patients with a pathological diagnosis of (thoracic) esophageal squamous cell carcinoma.
3. Age between 18 and 75 years (inclusive), both male and female.
4. Locally advanced esophageal squamous cell carcinoma without suspicious cervical lymph node metastasis and distant metastasis (cT1N1-3M0 or cT2-3N0-3M0, AJCC 8th edition).
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
6. No prior systemic treatment for esophageal cancer (including chemotherapy, targeted therapy, immune checkpoint inhibitors such as anti-PD-1 or PD-L1 antibodies, anti-CTLA-4 antibodies, etc.).
7. Planned surgical treatment after completion of neoadjuvant therapy.
8. Expected survival time of at least 6 months.
9. Clearly measurable lesions that meet the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
10. Adequate organ function based on laboratory values obtained during the screening period, including:

1) Hematology: no blood transfusions or blood products within 14 days, no use of G-CSF or other hematopoietic growth factors for correction, white blood cell count (WBC) ≥ 3.0 × 109/L, absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count (PLT) ≥ 75 × 109/L, hemoglobin (Hgb) ≥ 9 g/dL.

2) Blood chemistry: serum total bilirubin ≤ 1.5 × upper limit of normal (ULN), aspartate aminotransferase or alanine aminotransferase ≤ 2.5 × ULN (≤ 5 × ULN for patients with liver metastasis), serum creatinine ≤ 1.5 × ULN.

3) Coagulation function: prothrombin time (PT), international normalized ratio (INR) ≤ 1.5 × ULN.

4) Cardiac function: left ventricular ejection fraction (LVEF) ≥ 50%. 11. Female participants of childbearing potential must have a negative serum pregnancy test within 3 days before starting study drug and agree to use a medically accepted highly effective method of contraception (such as an intrauterine device, contraceptive pills, or condoms) during the study period and within 3 months after the last dose of study drug. Male participants with partners of childbearing potential must have undergone surgical sterilization or agree to use an effective method of contraception during the study period and within 3 months after the last dose of study drug.

Exclusion Criteria:

1. History of or concurrent active malignancy other than adequately treated non-melanoma skin cancer, curatively treated in situ cancer or other malignancy with no evidence of disease for at least 5 years.
2. Active bleeding within 3 months; a history of arterial or venous thrombotic events within 6 months, such as stroke (including transient ischemic attack), deep vein thrombosis, and pulmonary embolism; known inherited or acquired bleeding diathesis (e.g., coagulation factor deficiencies) or thrombotic disorders, such as patients with hemophilia; current or recent (within 10 days before the start of the study treatment) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes (allowed prophylactic use of low-dose aspirin and low-molecular-weight heparin); major surgery (excluding biopsy) within 4 weeks before starting study drug treatment or the surgical incision has not fully healed; current or recent (within 10 days before the start of the study treatment) use of aspirin (> 325 mg/day [maximum antiplatelet dose]) or other nonsteroidal anti-inflammatory drugs, dual antiplatelet therapy, clopidogrel, prasugrel, ticagrelor, or cilostazol.
3. The patient has received systemic treatment, surgery, or radiotherapy for esophageal cancer, including immunotherapy such as anti-PD-1 or PD-L1 antibodies, anti-CTLA-4 antibodies, targeted therapy, or chemotherapy.
4. The patient has used systemic corticosteroids or other systemic immunosuppressive drugs within 2 weeks before treatment, or is expected to use systemic immunosuppressive drugs during the trial. The use of inhaled glucocorticoids or physiological replacement doses of glucocorticoids is allowed.
5. The patient has active autoimmune diseases. Patients with type 1 diabetes, hypothyroidism requiring replacement therapy only, skin diseases (such as vitiligo, psoriasis, or alopecia) that do not require systemic treatment or are not expected to recur without external triggering factors can be included in the trial.
6. The patient has known active tuberculosis, is receiving anti-tuberculosis treatment, or has received anti-tuberculosis treatment within 1 year prior to the first dose.
7. The patient has severe, uncontrolled systemic diseases, such as refractory hypertension, severe active infection, etc.
8. The patient has known human immunodeficiency virus (HIV) infection or is known to be HIV-seropositive.
9. Untreated chronic hepatitis B or active carriers of hepatitis B virus (HBV) (HBV DNA >500 IU/mL) or active carriers of HCV detectable by HCV RNA. Note: Inactive carriers of hepatitis B surface antigen (HBsAg) or stable patients with treated chronic hepatitis B (HBV DNA < 500 IU/mL) can be included in the study.
10. History of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis, or symptomatic interstitial lung disease, or active pneumonia detected by chest CT scan within 4 weeks prior to initial drug treatment in the study.
11. Known symptomatic, untreated, or progressively advancing central nervous system (CNS) or leptomeningeal metastases.
12. Known allergy to any investigational drug or excipient.
13. Participation in other drug clinical trials within 4 weeks before enrollment.
14. Breastfeeding women.
15. As judged by the investigator, the patient has other factors that may affect the study results or may cause premature termination of the study, such as alcoholism, drug abuse, other serious illnesses (including mental illness) requiring concomitant treatment, significant laboratory abnormalities, or family or social factors that may affect the patient's safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response (pCR) of the patients' resected tumors | 1 month after resection
  PCR is defined as pT0N0M0

SECONDARY OUTCOMES:
Major pathologic response (MPR) | 1 month after resection
  MPR is defined as viable tumor comprised ≤ 10% of resected tumor specimens.
Disease Free Survival (DFS) | 3 and 5 years
  Percentage of Participants With DFS, as Assessed by RECIST 1.1. DFS is defined as the time from randomization to the first documented disease progression of local recurrence or distant metastasis or death due to any cause.
Overall Survival (OS) | 3 and 5 years
  OS is defined as the time from randomization to death due to any cause.
pathological downstaging rate | 1 month after resection
  The rate of patients with reduced pathological stage after neoadjuvant therapy
R0 resection rate | 1 month after resection
  The rate of patients with R0 resection after neoadjuvant therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Lulu Liu, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No